CLINICAL TRIAL: NCT05541432
Title: Finding the Optimal Resistance Training Intensity For Your Bones: A Randomized Controlled Trial (FORTIFY Bones)
Brief Title: Finding the Optimal Resistance Training Intensity For Your Bones
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Waterloo (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); University of Saskatchewan (Other); University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 41337
Record Dates: First submitted 2022-07-06; First posted 2022-09-15 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2024-05

CONDITIONS: Osteoporosis; Osteopenia
Keywords: Bone fracture; Strength training; Exercise; Bone mineral density; Muscle strength; Resistance training
MeSH Terms: conditions — Osteoporosis; Bone Diseases, Metabolic; Fractures, Bone; Motor Activity

STUDY DESIGN:
Intervention Model Description: Participants will be randomized in a 1:1:1 ratio to one of three arms. Participants will perform exercise or control activities twice weekly for 12 months. Not all participants will start and end at the same time.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Investigators and outcome assessors will be masked to the group allocation of participants. Participants will be masked to the hypothesis of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Home exercise (Active Comparator): Home exercise program, with biweekly group virtual education and exercise classes.
  Interventions: Other: Home exercise
- Supervised strength training (group 1) (Experimental): In-person, supervised muscle strengthening exercises twice weekly at a specific intensity.
  Interventions: Other: Supervised strength training (group 1)
- Supervised strength training (group 2) (Experimental): In-person, supervised muscle strengthening exercises twice weekly at a specific intensity.
  Interventions: Other: Supervised strength training (group 2)

INTERVENTIONS:
Other: Supervised strength training (group 1) — Participants in this arm will complete twice weekly resistance training. They will focus on form initially, and then be progressed to 3 sets of 10-12 repetitions at an intensity of ~70% of estimated 1 repetition maximum.
  Arms: Supervised strength training (group 1)
Other: Supervised strength training (group 2) — Participants in this arm will complete twice weekly resistance training. They will focus on form initially, and then be progressed to 3 sets of ~4-6 repetitions at an intensity of 85% of estimated one repetition maximum, with a warm-up set of 8 repetitions at their estimated 70% estimated one repetition maximum to attempt to match the volume performed in the other resistance training group.
  Arms: Supervised strength training (group 2)
Other: Home exercise — Participants in this arm will complete twice-weekly upper and lower body exercises at home, focused on posture and balance. Participants will meet 1:1 with an exercise physiologist who will select and prescribe exercises. Participants will also be invited to attend twice monthly virtual exercise and education sessions.
  Arms: Home exercise

SUMMARY:
Osteoporosis is a bone disease that can result in fractures, disability and an increased risk of premature death. Exercise is recommended for fall and fracture prevention, but health care professionals often recommend walking or lower intensity community exercise classes, which may not be effective for building bone. Further, individuals with osteoporosis are often told to avoid lifting or moving in certain ways, which creates fear and activity avoidance. Conversely, research suggests that to stimulate bone, you need higher loads on bone, with either higher intensity resistance training or impact exercise - the types of things people with low bone mass are told to avoid. Our study will examine different types of exercise intensity and how they translate to building bone in people with low bone mineral density (BMD).

DETAILED DESCRIPTION:
The FORTIFY Bones study will compare the effect of supervised twice-weekly progressive resistance training (PRT) at moderate or high intensity for one year to a home posture and balance exercise program on lumbar spine bone mineral density (BMD), in individuals with low bone mass not taking osteoporosis medication. As secondary analyses, we will examine the differences between each resistance training intensity and home exercise, and between resistance training intensities on all outcomes. Participants will be randomized to one of three exercise programs to be completed twice weekly: posture and balance exercise program at home, in-person, supervised progressive resistance training at 70% of estimated 1 Repetition Maximum (1RM) intensity, or in-person, supervised progressive resistance training at an 85% estimated 1RM intensity. The study is a multi-centre trial that will take place at the University of Waterloo, Toronto General Hospital, and the University of Saskatchewan. The long-term goal of this study is to generate evidence to support decision-making on the type of exercises for people with osteoporosis.

ELIGIBILITY:
Inclusion Criteria:

* Age 50 or over
* Has received 2 vaccines for COVID-19
* Has femoral neck, total hip, or lumbar spine BMD T-score of ≤ -1, OR has been or have a FRAX probability of fracture of greater than or equal to 20% for major osteoporotic fracture or 3% or greater for hip fracture.*

  * Individuals at high risk of fracture (i.e., risk in next 10 years is >20% according to FRAX) should be offered medication for osteoporosis. We will only include individuals at high risk of fracture who have declined medication or who had been on osteoporosis medication and decided to cease taking it in the appropriate timeline (as outlined by PI's and Physician).
* Willing to participate in 2x weekly exercise sessions
* Self-reported as postmenopausal for ≥ 2 years, OR postmenopausal stats confirmed via blood test (female participants only)

Exclusion Criteria:

* Is unable to communicate in English
* Has conditions affecting bone health
* Takes or has taken medications affecting bone in the last 12 months or longer (as determined by the research team)
* Has had a clinical or symptomatic spine fracture in the last 12 months, or a lower/upper limb fracture in the last 6 months
* Has had a joint replacement in the last 6 months
* Is receiving palliative care
* Has major surgery planned in the next 12 months
* Has had cancer within the last 2 years (excluding non-melanoma skin cancer)
* Has planned travel time of greater than 6 weeks
* Has been diagnosed with dementia
* Is already participating in moderate- or high-intensity progressive resistance training ≥ twice weekly
* Weighs over 450 lbs
* Has contraindications to resistance training

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 324 (Estimated)
Dates: Start 2022-09-13 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Lumbar Spine bone mineral density (BMD) | Baseline and 12 months
  Lumbar spine (L1-L4) bone mineral density measured via dual-energy X-ray Absorptiometry (DXA) scan.

SECONDARY OUTCOMES:
Fractures | Over 12 months
  Composite outcome of new non-vertebral and vertebral fractures, and progression of existing vertebral fractures. We will report the number in each category separately. We will use a fracture questionnaire for non-vertebral fractures, and vertebral fractures that come to clinical attention. Participants will undergo a DXA scan for Vertebral Fracture Assessment (VFA) at baseline and the 12-months. A vertebral fracture will be defined as having a radiographic presence of ≥25% reduction in anterior, middle, or posterior vertebral height, verified by an experienced radiologist at University Health Network via the Genant visual semi-quantitative method. Baseline VFA will be assessed for vertebral fractures and compared to VFA at 12 months to ascertain if there has been progression of new fractures; progression will be defined as progression to a new Genant level or a change in height of at least 10%.
Rate of falls per person per year | Over 12 months
  Participants will be emailed a falls calendar via a survey at the end of each month. Participants will be asked to immediately report any falls to research assistant and to exercise physiologist. Exercise physiologists will report any noted falls to their study coordinator immediately and additional follow-up documentation will be required. Rate of falls and number of people who experience one or more falls will be compared between groups.
Number of people who experience one or more falls | Over 12 months
  Participants will be emailed a falls calendar via a survey at the end of each month. Participants will be asked to immediately report any falls to research assistant and to exercise physiologist. Exercise physiologists will report any noted falls to their study coordinator immediately and additional follow-up documentation will be required. Rate of falls and number of people who experience one or more falls will be compared between groups.
Bone-free lean mass | Baseline and 12 months
  Whole body fat- and bone-free lean mass will be derived from DXA scans.
Appendicular lean mass | Baseline and 12 months
  We will calculate appendicular lean mass (kg) and its index (kg/m^2) from appendicular bone-free lean mass and height (cm).
Height | Baseline and 12 months
  Height will be a proxy measure of posture.
Occiput-to-wall distance | Baseline and 12 months
  Occiput-to-wall distance will be a proxy measure of posture.
Knee extension peak torque | Baseline, 6 months, and 12 months
  We will assess isometric knee extension peak torque using a knee extension test with a dynamometer.
30 Second Chair Stand Test. | Baseline, 6 months, and 12 months
  We will use the 30 Second Chair Stand Test.
Four Square Step Test | Baseline, 6 months, and 12 months
  We will use the Four Square Step Test to assess lower extremity muscle power and dynamic balance during functional tasks.
Grip Strength | Baseline, 6 months, and 12 months
  We will assess grip strength of the non-dominant arm using a hand dynamometer.
10 Metre Walk Test. | Baseline, 6 months, and 12 months
  We will assess gait speed using the 10 Metre Walk Test.
6 Minute Walk Test. | Baseline, 6 months, and 12 months
  We will assess endurance using the 6 Minute Walk Test.
Osteoporosis-specific quality of life (QUALEFFO-41) | Baseline, 6 months, and 12 months
  We will use the QUALEFFO-41 as an osteoporosis specific measure of health-related quality of life.
Quality of life (EQ5D5L) | Baseline, 6 months, and 12 months
  We will use the EQ5D5L measure as a generic health-related quality of life measure.
Serious adverse events | Over 12 months
  We will ask participants to report adverse events, using Health Canada definitions. We will report all serious and non-serious adverse events and identify those attributable to intervention. Safety outcomes will include all falls, fractures, and serious and non-serious adverse events. Any fractures or falls that are attributable to intervention will be considered under both fall or fracture outcomes, and harms.
Non-serious adverse events | Over 12 months
  We will ask participants to report adverse events, using Health Canada definitions. We will report all serious and non-serious adverse events and identify those attributable to intervention. Safety outcomes will include all falls, fractures, and serious and non-serious adverse events. Any fractures or falls that are attributable to intervention will be considered under both fall or fracture outcomes, and harms.
Glucose concentration | Baseline and 6 months
  We will be taking a fasted blood sample from participants to measure plasma glucose concentrations using biochemical assay. Blood samples will only be collected from participants at the University of Waterloo site.
Insulin concentration | Baseline and 6 months
  We will be taking a fasted blood sample from participants to measure serum insulin concentrations using radioimmunoassay. Blood samples will only be collected from participants at the University of Waterloo site.
Pro/anti-inflammatory markers | Baseline and 6 months
  We will be taking a fasted blood sample from participants to measure plasma pro- and anti-inflammatory markers using a multiplex kit. Blood samples will only be collected from participants at the University of Waterloo site.
Oxidative stress markers/antioxidant status (including oxygen radical absorbance capacity (ORAC) assay, protein carbonyls, glutathione peroxidase activity, thioredoxin, malondialdehyde) | Baseline and 6 months
  We will be taking a fasted blood sample from participants to measure antioxidant status and markers of oxidative stress using commercially available assays. Blood samples will only be collected from participants at the University of Waterloo site.
peptides synthesized and released by myocytes in muscle tissue | Baseline and 6 months
  We will be taking fasting blood samples from participants to measure peptides synthesized and released by myocytes in muscle tissue via the Luminex Performance Assay. Blood samples will only be collected from participants at the University of Waterloo site.
Total Hip BMD | Baseline and 12 months
  Bone mineral density of the hip measured via DXA scans
Femoral Neck BMD | Baseline and 12 months
  Bone mineral density of the femoral neck measured via DXA scans
Trabecular Bone Score | Baseline and 12 months
  Trabecular bone score (TBS) will be calculated using TBS iNsight software. A high TBS value indicates high quality boner structure, whereas a low TBS value demonstrates a lower quality structure. The TBS index ranges from 0.9 - 1.6.
Hip Geometry | Baseline and 12 months
  We will use the DXA scanner's hip structural analysis feature to calculate estimates of hip geometry from proximal femur scans.
Health Service Use | Baseline, 6 months, and 12 months
  We will assess direct medical resources (e.g., tests, medications, hospitalization, rehabilitation), direct non-medical resources (e.g., out of pocket expenses, transportation), indirect resources (e.g., iMTA Productivity Cost Questionnaire) and clinical events and management. We will assess resource use for incident falls, fractures or adverse events. Multiplying resources collected by jurisdictional unit costs in Canadian dollars will determine the total cost per exercise program.
Ratio of costs to QALY | Baseline, 6 months, and 12 months
  We will calculate the ratio of incremental costs between the interventions, determined by trial resources, and clinical outcome (QALY) to achieve an incremental cost per life year gained outcome.
Willingness to pay | Baseline, 6 months, and 12 months
  We will assess willingness to pay for various exercise models using a contingent valuation survey.
Body weight | Baseline, 6 months and 12 months
  Body weight in kg measured using scale

OTHER OUTCOMES:
Dietary Intake | Baseline, 6 months, and 12 months
  We will use Automated Self-Administered 24-hour dietary assessment tool (ASA24) to collect information on the participant's dietary intake through the self-administered 24-hour dietary record. Participants will report all food and beverage items and quantities on 3 days (2 weekday, 1 weekend day) at baseline, 6 months, and 12 months. We will also use the SCREEN2 tool at baseline only. We will report descriptive data on energy, protein, calcium, and vitamin D intake, and perform exploratory analyses of changes in these outcomes over time. We will perform subgroup analyses: 1) Baseline daily calcium (<1000 vs. >1000 mg per day); and 2) Baseline protein intake (<1.2g/kg body weight per day). We will explore changes in participants who are referred to a dietitian for counselling because of low intakes of protein, calcium, or vitamin D.

CONTACTS AND LOCATIONS:
Overall Officials: Lora Giangregorio, PhD, Principal Investigator — University of Waterloo
Locations (3):
- Canada (3):
  - University of Waterloo, Waterloo, Ontario
  - University of Toronto, Markham
  - University of Saskatchewan, Saskatoon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cauley JA, Thompson DE, Ensrud KC, Scott JC, Black D. Risk of mortality following clinical fractures. Osteoporos Int. 2000;11(7):556-61. doi: 10.1007/s001980070075. PMID 11069188
- [Background] Lindsay R, Silverman SL, Cooper C, Hanley DA, Barton I, Broy SB, Licata A, Benhamou L, Geusens P, Flowers K, Stracke H, Seeman E. Risk of new vertebral fracture in the year following a fracture. JAMA. 2001 Jan 17;285(3):320-3. doi: 10.1001/jama.285.3.320. PMID 11176842
- [Background] Ioannidis G, Papaioannou A, Hopman WM, Akhtar-Danesh N, Anastassiades T, Pickard L, Kennedy CC, Prior JC, Olszynski WP, Davison KS, Goltzman D, Thabane L, Gafni A, Papadimitropoulos EA, Brown JP, Josse RG, Hanley DA, Adachi JD. Relation between fractures and mortality: results from the Canadian Multicentre Osteoporosis Study. CMAJ. 2009 Sep 1;181(5):265-71. doi: 10.1503/cmaj.081720. Epub 2009 Aug 4. PMID 19654194
- [Background] Hopkins RB, Burke N, Von Keyserlingk C, Leslie WD, Morin SN, Adachi JD, Papaioannou A, Bessette L, Brown JP, Pericleous L, Tarride J. The current economic burden of illness of osteoporosis in Canada. Osteoporos Int. 2016 Oct;27(10):3023-32. doi: 10.1007/s00198-016-3631-6. Epub 2016 May 11. PMID 27166680
- [Background] Howe TE, Shea B, Dawson LJ, Downie F, Murray A, Ross C, Harbour RT, Caldwell LM, Creed G. Exercise for preventing and treating osteoporosis in postmenopausal women. Cochrane Database Syst Rev. 2011 Jul 6;2011(7):CD000333. doi: 10.1002/14651858.CD000333.pub2. PMID 21735380
- [Background] El-Khoury F, Cassou B, Charles MA, Dargent-Molina P. The effect of fall prevention exercise programmes on fall induced injuries in community dwelling older adults: systematic review and meta-analysis of randomised controlled trials. BMJ. 2013 Oct 29;347:f6234. doi: 10.1136/bmj.f6234. PMID 24169944
- [Background] Gillespie LD, Robertson MC, Gillespie WJ, Sherrington C, Gates S, Clemson LM, Lamb SE. Interventions for preventing falls in older people living in the community. Cochrane Database Syst Rev. 2012 Sep 12;2012(9):CD007146. doi: 10.1002/14651858.CD007146.pub3. PMID 22972103
- [Background] Sherrington C, Tiedemann A, Fairhall N, Close JC, Lord SR. Exercise to prevent falls in older adults: an updated meta-analysis and best practice recommendations. N S W Public Health Bull. 2011 Jun;22(3-4):78-83. doi: 10.1071/NB10056. PMID 21632004
- [Background] Tricco AC, Thomas SM, Veroniki AA, Hamid JS, Cogo E, Strifler L, Khan PA, Robson R, Sibley KM, MacDonald H, Riva JJ, Thavorn K, Wilson C, Holroyd-Leduc J, Kerr GD, Feldman F, Majumdar SR, Jaglal SB, Hui W, Straus SE. Comparisons of Interventions for Preventing Falls in Older Adults: A Systematic Review and Meta-analysis. JAMA. 2017 Nov 7;318(17):1687-1699. doi: 10.1001/jama.2017.15006. PMID 29114830
- [Background] Duckham RL, Masud T, Taylor R, Kendrick D, Carpenter H, Iliffe S, Morris R, Gage H, Skelton DA, Dinan-Young S, Brooke-Wavell K. Randomised controlled trial of the effectiveness of community group and home-based falls prevention exercise programmes on bone health in older people: the ProAct65+ bone study. Age Ageing. 2015 Jul;44(4):573-9. doi: 10.1093/ageing/afv055. Epub 2015 Apr 23. PMID 25906791
- [Background] Nikander R, Gagnon C, Dunstan DW, Magliano DJ, Ebeling PR, Lu ZX, Zimmet PZ, Shaw JE, Daly RM. Frequent walking, but not total physical activity, is associated with increased fracture incidence: a 5-year follow-up of an Australian population-based prospective study (AusDiab). J Bone Miner Res. 2011 Jul;26(7):1638-47. doi: 10.1002/jbmr.363. PMID 21328475
- [Background] Rikkonen T, Salovaara K, Sirola J, Karkkainen M, Tuppurainen M, Jurvelin J, Honkanen R, Alhava E, Kroger H. Physical activity slows femoral bone loss but promotes wrist fractures in postmenopausal women: a 15-year follow-up of the OSTPRE study. J Bone Miner Res. 2010 Nov;25(11):2332-40. doi: 10.1002/jbmr.143. PMID 20533310
- [Background] Sherrington C, Fairhall NJ, Wallbank GK, Tiedemann A, Michaleff ZA, Howard K, Clemson L, Hopewell S, Lamb SE. Exercise for preventing falls in older people living in the community. Cochrane Database Syst Rev. 2019 Jan 31;1(1):CD012424. doi: 10.1002/14651858.CD012424.pub2. PMID 30703272
- [Background] Costa AG, Wyman A, Siris ES, Watts NB, Silverman S, Saag KG, Roux C, Rossini M, Pfeilschifter J, Nieves JW, Netelenbos JC, March L, LaCroix AZ, Hooven FH, Greenspan SL, Gehlbach SH, Diez-Perez A, Cooper C, Compston JE, Chapurlat RD, Boonen S, Anderson FA Jr, Adachi JD, Adami S. When, where and how osteoporosis-associated fractures occur: an analysis from the Global Longitudinal Study of Osteoporosis in Women (GLOW). PLoS One. 2013 Dec 11;8(12):e83306. doi: 10.1371/journal.pone.0083306. eCollection 2013. PMID 24349484